CLINICAL TRIAL: NCT02919501
Title: Interventional, Randomised, Double-blind, Parallel-group Study of the Efficacy and Safety of Initial Administration of 17 mg Vortioxetine Intravenously With 10 mg/Day Vortioxetine Orally in Patients With Major Depressive Disorder
Brief Title: Study of the Efficacy and Safety of Initial Administration of 17 mg Vortioxetine Intravenously With 10 mg/Day Vortioxetine Orally in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16903A; 2015-005081-30 (EudraCT Number)
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine (IV); Drug: Vortioxetine (tablet)
- IV placebo (Placebo Comparator)
  Interventions: Other: Placebo (IV); Drug: Vortioxetine (tablet)

INTERVENTIONS:
Drug: Vortioxetine (IV) — 17 mg, solution for infusion, administered, over 2 hours as single dose
  Arms: IV vortioxetine
Other: Placebo (IV) — Saline: isotonic sodium chloride, administered, over 2 hours as single dose
  Arms: IV placebo
Drug: Vortioxetine (tablet) — 10 mg, tablets, oral administration once daily for 15 days (open labelled)

SUMMARY:
To evaluate the early onset of efficacy of vortioxetine 17 mg intravenously (IV) and vortioxetine 10 mg/day oral dose regimen versus placebo IV and vortioxetine 10 mg/day oral dose regimen on depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

* The patient has recurrent Major Depressive Disorder (MDD), diagnosed according to Diagnostic and Statistical Manual for Mental Disorders, 5th Edition (DSM-5™), classification code (296.3x). The recurrent Major Depressive Episode (MDE) should be confirmed using the Mini-International Neuropsychiatric Interview (MINI).
* The patient has a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≥30 at both Screening and Baseline Visits.
* The patient has had the current MDE for ≥3 months

Exclusion Criteria:

* The patient has any current psychiatric disorder or Axis I disorder (DSM-5™ criteria), other than MDD, as assessed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has a current diagnosis of history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features (DSM-5™ criteria).
* The patient suffers from personality disorders, intellectual disability, pervasive development disorder, attention deficit/hyperactivity disorder, organic mental disorders, or mental disorders due to a general medical condition (DSM-5™ criteria).
* The patient has a history of lack of response to previous treatment with vortioxetine (including current episode).

Other Protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 1 in MADRS total score | Baseline to Week 1
  The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.

SECONDARY OUTCOMES:
Change from baseline to Week 2 in MADRS total score | Baseline to Week 2
  The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Change from baseline to Day 3 in MADRS total score | Baseline to Day 3
  The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Change from baseline to Day 1 in MADRS total score | Baseline to Day 1
  The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Response (defined as a ≥ 50% decrease in MADRS total score from baseline) at Week 1 | Week 1
Remission at Week 1 (defined as a MADRS total score ≤ 10) | Week 1
Change from baseline to Week 1 in HADS depression subscale | baseline to Week 1
  The Hospital Anxiety and Depression Scale (HADS) is a patient-rated scale designed to screen for anxiety and depressive states in medical patients. It consists of two sub-scales: the D-scale measures depression and the A-scale measures anxiety. Each sub-scale contains 7 items, and each item is rated from 0 (absent) to 3 (maximum severity). The score of each sub-scale ranges from 0 to 21.
Global clinical impression -Global Improvement | At Week 1
  The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Change from baseline in Global clinical impression -Severity | Baseline to Week 1
  The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients
Oral clearance (CL/F) | 2, 8 and 24 hours postdose (day 1) and day 14
Average Plasma Concentration (Cav) | 2, 8 and 24 hours postdose (day 1) and day 14
Change from baseline to Week 1 in HADS anxiety subscale | Baseline to Week 1
  The HADS is a patient-rated scale designed to screen for anxiety and depressive states in medical patients. It consists of two sub-scales: the D-scale measures depression and the A-scale measures anxiety. Each sub-scale contains 7 items, and each item is rated from 0 (absent) to 3 (maximum severity). The score of each sub-scale ranges from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (7):
- Estonia (2):
  - EE1019, Tallinn
  - EE1020, Tallinn
- Finland (5):
  - FI1040, Helsinki
  - FI1041, Helsinki
  - FI1030, Kuopio
  - FI1009, Pori
  - FI1027, Turku

REFERENCES:
- [Derived] Vieta E, Florea I, Schmidt SN, Areberg J, Ettrup A. Intravenous vortioxetine to accelerate onset of effect in major depressive disorder: a 2-week, randomized, double-blind, placebo-controlled study. Int Clin Psychopharmacol. 2019 Jul;34(4):153-160. doi: 10.1097/YIC.0000000000000271. PMID 31094901
- See also: Results EudraCT 2015-005081-30 — http://www.clinicaltrialsregister.eu/ctr-search/trial/2015-005081-30/results